CLINICAL TRIAL: NCT01740596
Title: C-Pulse Heart Assist Device pivOtal stUdy treatiNg paTients With modERate to Severe Heart Failure C-Pulse® System: A Heart Assist Device Pivotal IDE Study
Brief Title: C-Pulse® System: A Heart Assist Device Clinical Study
Acronym: COUNTER-HF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped early due to a business decision to no longer pursue commercialization of the C-PULSE System. This decision was not based on any safety concerns.
Sponsor: Nuwellis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO 03970-C
Record Dates: First submitted 2012-11-28; First posted 2012-12-04 (Estimated); Results first posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-08

CONDITIONS: Heart Failure
Keywords: NYHA III; NYHA IV; ACC Stage C; Heart Failure; Congestive Heart Failure; C-Pulse; Counterpulsation; Heart Assist; Sunshine Heart; Left Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- C-Pulse® System (Experimental): C-Pulse® System Counterpulsation
  Interventions: Device: C-Pulse® System Counterpulsation
- Control Arm (No Intervention): Optimal Medical Therapy

INTERVENTIONS:
Device: C-Pulse® System Counterpulsation — The Sunshine Heart C-Pulse System is an implantable, non-blood contacting, non-obligatory, heart assist device. The system provides cardiac assistance through an extra-aortic balloon Cuff and ECG sense lead connected by means of a Percutaneous Interface Lead (PIL) to an external pneumatic Driver. The PIL is held secure externally, at the exit site, with a simple adhesive clip (C-Patch or similar) for immobilization of the external part of the PIL. The Driver is adjusted using a dedicated notebook computer (Programmer) with specialized software.
  Arms: C-Pulse® System

SUMMARY:
Sunshine Heart is sponsoring a prospective, multi-center, randomized trial to assess the safety and efficacy of the C-Pulse® System ("C-Pulse").

The purpose of the study is to determine whether the use of the C-Pulse as a treatment for patients in moderate to severe heart failure (HF) has demonstrated safety and efficacy, such that the C-Pulse System merits Food and Drug Administration (FDA) approval to market the device in the United States.

DETAILED DESCRIPTION:
The C-Pulse® System is indicated for use in patients with moderate to severe heart failure while on optimal heart failure drug and on device therapies. The C-Pulse® System is intended to relieve the symptoms of heart failure, improve quality of life and cardiac function, and reduce the need for heart failure hospitalization. It is intended for use in hospital and at home. It is not intended as a replacement for heart function; it is not life sustaining or life-supporting therapy. It does not preclude the use of other heart failure therapies, such as valve surgery, heart transplantation or LVAD.

The Sunshine Heart C-Pulse System is an implantable, non-blood contacting, non-obligatory, heart assist device. The system provides cardiac assistance through an extra-aortic balloon Cuff and ECG sense lead connected by means of a Percutaneous Interface Lead (PIL) to an external pneumatic Driver. The PIL is held secure externally, at the exit site, with a simple adhesive clip (C-Patch or similar) for immobilization of the external part of the PIL. The Driver is adjusted using a dedicated notebook computer (Programmer) with specialized software.

The non-blood contacting feature of the C-Pulse® System also allows the device to be intermittently turned off as tolerated. This allows the patient freedom for personal hygiene.

ELIGIBILITY:
Inclusion Criteria:

1. Left ventricular ejection fraction (LVEF) ≤ 35% (by transthoracic ECHO within 90 days prior to randomization)
2. ACC/AHA Stage C and NYHA III to ambulatory Class IV
3. Age ≥ 18 years
4. Must have cardiac resynchronization therapy (CRT) when clinically indicated, implanted ≥90 days prior to randomization.
5. Must have an implanted cardio-defibrillator (ICD) when clinically indicated, implanted at least 30 days prior to randomization.

   Note: If a subject is clinically indicated for an ICD but refuses the ICD, he/she may be enrolled. Please document the refusal of the ICD in the medical record and the eCRFs.
6. Patient must be on stable, up-titrated medical therapy as recommended according to current guidelines (Circulation. 2009; 119 (12): 1977-2016) which minimally includes:

   * ACE-inhibitor (ACE-I) at stable doses for 1 month prior to enrollment, if tolerated, AND
   * a beta blocker (carvedilol, sustained release metoprolol succinate, or bisoprolol) for 3 months prior to enrollment, if tolerated, with a stable up-titrated dose for 1 month prior to enrollment.
   * This also includes an Angiotensin II Receptor Blocker (ARB) at stable doses for 1 month prior to enrollment, if tolerated, when ACE-I is not tolerated.
   * Stable is defined as no more than a 100% increase or a 50% decrease in dose. If the patient is intolerant to ACE-I, ARB, or beta blockers, documented evidence must be available.
   * In those intolerant to both ACE-I and ARB, combination therapy with hydralazine and oral nitrate should be considered. Therapeutic equivalence for ACE-I substitutions is allowed within the enrollment stability timelines.
   * Aldosterone inhibitor therapy should be added. Eplerenone requires dosage stability for 1 month prior to enrollment.
   * Diuretics may be used as necessary to keep the patient euvolemic.
7. Functional limitation due to heart failure as defined by a 6 Minute Walk test of ≥ 175 ≤ 375 meters, measured within 30 days prior to randomization
8. At least one hospitalization for decompensated heart failure as defined below, while on heart failure medications, within 12 months prior to randomization or BNP level > 300 or NTproBNP > 1500

   Heart failure related hospitalization is defined by the following:
   * signs and symptoms of worsening heart failure; and
   * treatment with intravenous heart failure therapy (including but not limited to diuretic or inotropic therapy) and
   * a minimum of one date change in the hospital
9. Patient understands the nature of the procedure and on-going device therapy, is willing to comply with associated follow-up evaluations, and provide written informed consent prior to the procedure.

Exclusion Criteria:

1. Any evidence, as assessed within 90 days prior to enrollment, of either:

   1. Ascending aortic calcification on posterior-anterior or lateral chest x-ray
   2. Calcific ascending aortic disease as detected by non-contrast CT scan
   3. Ascending aorto-coronary artery bypass grafts, history of aortic dissection, Marfans disease or other connective tissue disorder or repaired aortic coarctation OR
   4. Has had an ascending aortic composite graft or root replacement
2. Aorta not conforming to specified dimensional constraints defined by CT scan, most specifically mid ascending aortic outside diameter less than 28 mm or greater than 42 mm
3. Inotrope dependence - inability to wean from inotropic therapy
4. ACC/AHA Stage D heart failure or non-ambulatory NYHA Class IV subject
5. Hypertrophic obstructive cardiomyopathy, restrictive cardiomyopathy, pericardial disease, amyloidosis, active myocarditis, diastolic heart failure or technically challenging congenital heart disease
6. Reversible cause of heart failure that may be remedied by conventional surgery or other intervention
7. Moderate to severe aortic insufficiency (≥ 2+)
8. ST elevation myocardial infarction (STEMI) within 30 days prior to randomization
9. Cardiac surgery within 90 days prior to randomization
10. Prior cardiac transplantation, left ventricular reduction surgery, passive restraint device or surgically implanted left ventricular assist device
11. Anticipated concomitant cardiac surgical procedure
12. Serum creatinine ≥ 2.5mg/dL or any form of dialysis within 30 days prior to randomization
13. Evidence of intrinsic hepatic disease as defined as biopsy proven liver cirrhosis; or liver enzyme values (AST, ALT or total bilirubin) that are > 3 times the upper limit of normal within 30 days prior to randomization
14. Patient has severe intrinsic pulmonary disease in judgment of the investigator
15. Body Mass Index (BMI) < 18 or > 45 kg/m2
16. Suspected or active systemic infection

    1. Within 14 days prior to randomization and
    2. Evidenced by positive culture, antibiotics for empiric treatment or elevated WBC > 12K and temperature >38o C
17. Stroke or transient ischemic attack (TIA) within the 90 days prior to randomization; or > 80% carotid stenosis as determined by carotid Doppler ultrasound within 90 days prior to randomization
18. Positive serum pregnancy test, for women of childbearing potential
19. Patient has a condition, other than heart failure, which would limit survival to less than 2 years
20. Patient is currently enrolled or has participated in the last 30 days in another therapeutic or interventional clinical study
21. Patient demonstrates compliance issues that in the opinion of the investigator could interfere with the ability to manage the therapy (i.e. uncontrolled diabetes, mental health issues, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-09-12 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Abraham, MD, Principal Investigator — Ohio State University; Margarita T Camacho, MD, Principal Investigator — Newark Beth Israel
Locations (28):
- United States (28):
  - The University of Alabama at Birmingham Hospital, Birmingham, Alabama
  - University of Southern California Keck School of Medicine, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Morton Plant Hospital, Clearwater, Florida
  - Memorial Healthcare System, Hollywood, Florida
  - University of Miami Medical Center, Miami, Florida
  - Medical Center of Central Georgia, Macon, Georgia
  - University of Louisville - Jewish Hospital, Louisville, Kentucky
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Mid America Heart Institute-Saint Luke's Hospital, Kansas City, Missouri
  - St. Louis Heart and Vascular, St Louis, Missouri
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Cornell University, New York - Presbyterian Hospital, New York, New York
  - Westchester Medical Center, Valhalla, New York
  - Charlotte-Mecklenburg Hospital - Carolinas Health Care System, Charlotte, North Carolina
  - The Ohio State University Medical Center, Columbus, Ohio
  - Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Allegheny-Singer Research Institute - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Dallas VA Medical Center, Dallas, Texas
  - Texas Heart Institute - St Luke's Hospital, Houston, Texas
  - VCU Medical Center, Richmond, Virginia
  - Providence Sacred Heart Medical Center, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Implants
Groups:
- C-Pulse® System Treatment Group: C-Pulse® System Counterpulsation: The Sunshine Heart C-Pulse System is an implantable, non-blood contacting, non-obligatory, heart assist device. The system provides cardiac assistance through an extra-aortic balloon Cuff and ECG sense lead connected by means of a Percutaneous Interface Lead (PIL) to an external pneumatic Driver. The PIL is held secure externally, at the exit site, with a simple adhesive clip (C-Patch or similar) for immobilization of the external part of the PIL. The Driver is adjusted using a dedicated notebook computer (Programmer) with specialized software.
  + Continued Optimal Medical Therapy.
- Control Group: Continued Optimal Medical Therapy
Period: Overall Study
Arm/Group | C-Pulse® System Treatment Group | Control Group
Started | 19; 16 Implants | 19; 0 Implants
Completed | 0; 0 Implants | 0; 0 Implants
Not Completed | 19; 16 Implants | 19; 0 Implants

BASELINE CHARACTERISTICS:
Population: Study was closed early with only 38/388 (9.8%) subjects enrolled and Baseline Characteristics were analyzed collectively across both treatment arms of the study. A total of 38 patients were randomized, however, 3/38 patients randomized to the Treatment Arm were withdrawn from the study prior to implant occurring and were not included in the final analysis. The overall number of baseline participants analyzed was 35/38.
Groups:
- Study Participants: Study participants consisted of Treatment Arm (n=17) who received the C-Pulse System and Control Arm (n=18) who received standard optimal medical therapy.
Arm/Group | Study Participants
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] — Age Range: 42.0-78.0 years Population: There were 35 subjects analyzed in total with 17 in treatment arm and 18 in control.
  years
    Treatment Arm: number analyzed (Participants) | 17
    Treatment Arm | 63.3 (11.7)
    Control Arm: number analyzed (Participants) | 18
    Control Arm | 58.5 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: There were 35 subjects analyzed in total with 17 in treatment arm and 18 in control.
  Participants
    Treatment Arm: number analyzed (Participants) | 17
    Treatment Arm: Female | 2
    Treatment Arm: Male | 15
    Control Arm: number analyzed (Participants) | 18
    Control Arm: Female | 4
    Control Arm: Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: There were 35 subjects analyzed in total with 17 in treatment arm and 18 in control.
  Participants
    Treatment Arm: number analyzed (Participants) | 17
    Treatment Arm: Black or African American | 5
    Treatment Arm: Caucasian | 9
    Treatment Arm: Not Disclosed | 3
    Control Arm: number analyzed (Participants) | 18
    Control Arm: Black or African American | 8
    Control Arm: Caucasian | 9
    Control Arm: Not Disclosed | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35
Intermacs Subject Profile/Status [Count of Participants; unit: Participants] — INTERMACS provide prognostic information for patients with advanced heart failure receiving mechanical support Population: There were 35 subjects analyzed in total with 17 in treatment arm and 18 in control.
  Participants
    Treatment Arm: number analyzed (Participants) | 17
    Treatment Arm: 4: Resting Symptoms | 0
    Treatment Arm: 5: Exertion Intolerant | 6
    Treatment Arm: 6: Exertion Limited | 7
    Treatment Arm: 7: Advanced NYHA Class III | 3
    Treatment Arm: Not Available | 1
    Control Arm: number analyzed (Participants) | 18
    Control Arm: 4: Resting Symptoms | 4
    Control Arm: 5: Exertion Intolerant | 3
    Control Arm: 6: Exertion Limited | 7
    Control Arm: 7: Advanced NYHA Class III | 1
    Control Arm: Not Available | 3
NYHA Classification [Count of Participants; unit: Participants] — NYHA class defines limitation of physical activity I: No limitation II: Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  III: Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  IV: Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases. Population: There were 35 subjects analyzed in total with 17 in treatment arm and 18 in control.
  Participants
    Treatment Arm: number analyzed (Participants) | 17
    Treatment Arm: Class I | 0
    Treatment Arm: Class II | 0
    Treatment Arm: Class III | 17
    Treatment Arm: Class IV | 0
    Control Arm: number analyzed (Participants) | 18
    Control Arm: Class I | 0
    Control Arm: Class II | 0
    Control Arm: Class III | 18
    Control Arm: Class IV | 0

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Outcome
Description: The primary safety endpoint is serious procedure and device related adverse events as determined by CEC adjudication. No formal statistical hypotheses.
Time Frame: 4 Years Follow-up
Population: Study was closed early with only 38 randomized subjects (19 treatment group and 19 control). Primary and secondary endpoints were not statistically evaluated as there was insufficient sample size and follow-up. The primary safety outcome was only applicable to the implant treatment arm as it is specifically measuring device and/or procedure related serious adverse events (control arm was treated as standard of care and did not undergo a procedure for the study device to be placed).
Measure: Count of Participants; unit: Participants
Groups:
- Study Participants: C-Pulse® System Treatment Group
Arm/Group | Study Participants
Number analyzed (Participants) | 19
Participants
  Device Related Serious Adverse Event (infection, device malfunction, worsening heart failure) | 5
  Procedure Related Serious Adverse Events (MI, arrhythmias, fluid collection) | 6

2. Secondary Outcome: Improvement in 6 Minute Hall Walk (6MW) at 12-months
Description: improvement of distance walked during the 6MW at 12-months.
Time Frame: 12-months
Population: Number of participants that completed the 6MW
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | C-Pulse® System Treatment Group | Control Group
Number analyzed (Participants) | 4 | 10
meters | 279 (164) | 289 (95)

3. Secondary Outcome: Improvement in LVEF at 12 Months.
Description: Improvement in left ventricular ejection fraction (LVEF) at 12 months.
Time Frame: 12-months
Population: Number of participants with LVEF at 12-months.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | C-Pulse® System Treatment Group | Control Group
Number analyzed (Participants) | 5 | 8
percentage | 22.0 (2.7) | 22.0 (7.6)

4. Secondary Outcome: Improvement in KCCQ Score at 12-months.
Description: The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a quality-of-life assessment for heart failure patients taking into consideration severity of heart failure symptoms and limitations patients experience. The scores are scaled from 0 to 100 and frequently summarized in 25-point ranges, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent
Time Frame: 12-months
Population: Number of Participants that completed the KCCQ at 12-months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | C-Pulse® System Treatment Group | Control Group
Number analyzed (Participants) | 5 | 9
score on a scale | 61.4 (23.1) | 52.3 (22.5)

ADVERSE EVENTS:
Time Frame: Up to 4 years of follow-up.
Groups:
- Treatment Group: C-Pulse® System Treatment group
Arm/Group | Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 10/19 | 5/19
Serious Adverse Events (participants affected / at risk) | 16/19 | 15/19
Other Adverse Events (participants affected / at risk) | 9/19 | 1/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=19) | Control Group (N=19)
Major Infection (Infections and infestations) | 6 (13) | 3 (4) — Major infection: localized non-device, percutaneous site and/or pocket, or sepsis
Cardiac Disorders (Cardiac disorders) | 11 (21) | 10 (10) — Cardiac arrhythmias, myocardial infarction, pericardial fluid collection
Worsening Heart Failure (Cardiac disorders) | 13 (28) | 13 (24)
Renal or Neuro Dysfunction (General disorders) | 8 (18) | 5 (7)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Device Malfunction (Product Issues) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=19) | Control Group (N=19)
Cardiac Disorders (Cardiac disorders) | 4 (4) | 0 (0) — Cardiac arrhythmias, bleeding
General Disorders (General disorders) | 4 (5) | 1 (4) — Hepatic dysfunction
Infection (Infections and infestations) | 4 (5) | 0 (0) — Infection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-08-14): https://cdn.clinicaltrials.gov/large-docs/96/NCT01740596/Prot_SAP_ICF_000.pdf